CLINICAL TRIAL: NCT02969330
Title: Effect of Short Peripheral Electrical Stimulation (PES) on Brain Response to Glucose Stimuli Evaluated by BOLD and Functional Diffusion MRI: a Crossover Pilot Study
Brief Title: Effect of Peripheral Electrical Stimulation (PES) on Brain Response to Glucose Stimuli
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel Aviv University (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Uri Nevo, PhD, Tel Aviv University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2366-16-SMC
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Brain Activity; Glucose Control
MeSH Terms: interventions — Tissue Therapy, Historical; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose (Experimental): Glucose ingestion
  Interventions: Dietary Supplement: Glucose
- PES (Active Comparator): Single session of short PES treatment before glucose ingestion.
  Interventions: Device: Stimulator; Dietary Supplement: Glucose

INTERVENTIONS:
Device: Stimulator
  Arms: PES
Dietary Supplement: Glucose — 300ml tap water with 75g glucose

SUMMARY:
The aims of this study are twofold: (1) to develop an innovative approach for studying brain glucose metabolism using functional diffusion weighted imaging (DWI) and BOLD fMRI in humans; (2) to evaluate the effect of short peripheral electrical stimulation (PES) treatment on brain and brain-stem targets, associated with control of food intake and energy expenditure, in response to glucose stimuli, in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 18-65 years old.
* Body mass index 18 to 25 kg/m2
* Capable of giving informed consent

Exclusion Criteria:

* Pregnancy, or nursing
* Permanent pacemakers
* Metal prosthesis
* Skin disease
* Claustrophobia
* History of neurological disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Changes in postprandial cerebral blood flow (fMRI) and cerebral diffusivity (fDWI) in response to glucose ingestion. | changes from baseline to 30 minutes after glucose ingestion

IPD SHARING:
Plan to Share IPD: No